CLINICAL TRIAL: NCT01065792
Title: Re-examination Study for General Drug Use to Assess the Safety and Efficacy Profile of STOCRIN in Usual Practice
Brief Title: Stocrin Re-examination Study (0831-028)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 0831-028; 2010_008 (Other: Merck)
Record Dates: First submitted 2010-02-08; First posted 2010-02-09 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: HIV Infection
Keywords: HIV Infection
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients with HIV-1 infection taking Stocrin

SUMMARY:
This survey is conducted for preparing application materials for re-examination under the Pharmaceutical Affairs Laws and its Enforcement Regulation, its aim is to reconfirm the clinical usefulness of STOCRIN through collecting the safety and efficacy information according to the Re-examination Regulation for New Drugs.

Post-marketing surveys are not considered applicable clinical trials and thus the results of this survey will not be posted at its conclusion. The results will be submitted to public health officials as required by applicable national and international laws.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 Infected Patient
* Patient Who Is Treated With Stocrin 600 Mg Tablet Within Local Label During The Enrollment Period (A Patient Who Changes The Therapy From Stocrin 200 Mg Capsule To Stocrin 600 Mg Tablet Can Be Eligible.)

Exclusion Criteria:

* Patient Who Has A Contraindication To Stocrin According To The Local Label

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with HIV-1 infection treated with STOCRIN
Sampling Method: Probability Sample
Enrollment: 728 (Actual)
Dates: Start 2009-03; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Percent of patients with any adverse experience | Up to 14 days following cessation of treatment
Proportion of patients with HIV-1 RNA levels of less than 400 copies per milliliter after treatment | At 12 weeks +/- 2 weeks and at 24 weeks +/- 2 weeks after first treatment
Change from baseline in CD4 cell count and overall efficacy evaluation by investigator (success, failure or can not be assessed) | At 12 weeks +/- 2 weeks and at 24 weeks +/- 2 weeks after first treatment

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC